CLINICAL TRIAL: NCT03238014
Title: Efficacy of High-intensity Noninvasive Positive Pressure Ventilation and Low-intensity Noninvasive Positive Pressure Ventilation in Patients With Chronic Hypercapnic Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy of High-intensity NPPV and Low-intensity NPPV in Patients With Chronic Hypercapnic COPD
Acronym: NPPV;COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guan Lili, Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GIRD201707
Record Dates: First submitted 2017-07-27; First posted 2017-08-03 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: COPD; Hypercapnic Respiratory Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity noninvasive ventilation (Experimental): High-intensity noninvasive positive pressure ventilation aims at maximally improving PaCO2.
  Interventions: Device: Noninvasive positive pressure ventilation
- Low-intensity noninvasive ventilation (Active Comparator): Low-intensity noninvasive positive pressure ventilation is a classic setting of noninvasive ventilation.
  Interventions: Device: Noninvasive positive pressure ventilation

INTERVENTIONS:
Device: Noninvasive positive pressure ventilation — Noninvasive positive pressure ventilation used assist/control mode treat severe stable chronic obstructive pulmonary disease.
  Other Names: Noninvasive ventilation

SUMMARY:
High-intensity noninvasive positive pressure ventilation (NPPV), which can well improve the gas exchange and reduce the work of breathing of patients, is a new strategy targeted at maximally reducing arterial carbon dioxide. However, no definitive conclusions have been drawn to decide whether high-intensity NPPV is the best setting for treating patients with chronic hypercapnic COPD. For now, no unified method for setting up high-pressure NPPV has been established. Most of the trials utilized gradually increased inspiratory positive airway pressure depending on the patient's tolerance. However, from a respiratory physiology point of view, excessive inspiratory positive airway pressure may lead to lung hyperinflation, increased intrinsic positive end expiratory pressures, increased oxygen consumption, and ineffective work of breathing.Therefore, seeking a method to establish individualized high-intensity NPPV is of vital importance.

ELIGIBILITY:
Inclusion Criteria:

Clinically stable with chronic hypercapnic COPD (baseline arterial carbon dioxide pressure (PaCO2) of 50 mmHg or higher, measured resting in a sitting position and breathing room air without having used NPPV for at least 1 hour)

Exclusion Criteria:

* other lung/pleural diseases or thoracic deformity
* severe heart failure (New York Heart Association class IV), severe dysrhythmia
* unstable angina, or malignant comorbidity
* obesity (BMI ≥ 35 kg/m²)
* severe obstructive sleep apnea syndrome

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Partial pressure of arterial blood carbon dioxide (PaCO2) | 12 weeks
  Daytime arterial blood gas samples were taken with patients resting in a sitting position and breathing room air without having used NPPV for at least 1 hour.

SECONDARY OUTCOMES:
Severe Respiratory Insufficiency (SRI) Questionnaire | 12 weeks
  The SRI Questionnaire has good psychometric properties shown to be valid for chronic hypercapnic COPD patients receiving NPPV. It includes 49 items on seven subscales.
Baseline Dyspnea Index/Transition Dyspnea Index | 12 weeks
  Baseline Dyspnea Index/Transition Dyspnea Index provides a multidimensional measurement of dyspnea based on 3 components that evoke dyspnea in activities of daily living, in symptomatic individuals.
Chromic Respiratory Questionnaire | 12 weeks
  Chromic Respiratory Questionnaire is uesd to measure the health related quality of life in patients with chronic respiratory disease.
COPD assessment test | 12 weeks
  The COPD Assessment Test is a questionnaire for people with COPD. It is designed to measure the impact of COPD on a person's life, and how this changes over time.
Pulmonary function | 12 weeks
  Pulmonary function tests of lung mechanics - measurements of forced vital capacity, forced expiratory volume in 1 second, forced inspiratory flow rates, etc.
6-minute walk test | 12 weeks
  The 6-minute walk test plays a key role in evaluating functional exercise capacity, assessing prognosis and evaluating response to treatment across a wide range of respiratory diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, Study Director — Guangzhou Institute of Respiratory Disease
Locations (1):
- Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong, China